CLINICAL TRIAL: NCT03430037
Title: AFFIRM: A Phase 2 Randomized, Placebo-Controlled Study of Alleviation by Fisetin of Frailty, Inflammation, and Related Measures in Older Women
Brief Title: Alleviation by Fisetin of Frailty, Inflammation, and Related Measures in Older Women
Acronym: AFFIRM
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert J. Pignolo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-000472
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Frail Elderly Syndrome
Keywords: Inflammation; Frailty
MeSH Terms: conditions — Inflammation; Frailty | interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Fisetin 20/mg/kg/day, orally for 2 consecutive days, for 2 consecutive months.
  Interventions: Dietary Supplement: Fisetin
- Placebo (Placebo Comparator): Placebo capsules orally for 2 consecutive days, for 2 consecutive months.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Dietary Supplement: Fisetin — Flavonoid Family
  Arms: Treatment
Drug: Placebo oral capsule — Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a pilot study to evaluate whether targeting inflammation will help reduce markers of insulin resistance inflammation, bone resorption and physical dysfunction in elderly women with gait disturbance. Positive results of this study would lead to the development of a larger clinical trial examining the effects of this intervention on age-related dysfunction.

DETAILED DESCRIPTION:
To the researchers' knowledge, there are no published studies utilizing Fisetin in alteration of frailty markers. Several studies involve use of Fisetin for its anti-oxidative and anti-apoptotic effects in animal models. Fisetin may reduce oxidative stress, alleviate hyperglycemia, and improve kidney function. No one has evaluated the biologic markers of inflammation and frailty in older postmenopausal women. The researchers plan to evaluate markers of frailty and markers of inflammation, insulin resistance, and bone resorption while maintaining bone formation in older postmenopausal women.

ELIGIBILITY:
Inclusion Criteria

* Healthy postmenopausal women
* Age ≥ 70 years

Exclusion Criteria

* Abnormality in any of the screening laboratory studies (see below)
* Presence of significant liver or renal disease
* Malignancy (including myeloma)
* Malabsorption
* Hypoparathyroidism
* Hyperparathyroidism
* Acromegaly
* Cushing's syndrome
* Hypopituitarism
* Gastric bypass/reduction
* Malabsorption issues
* Crohn's
* Myopathies (increased or low calcium, vitamin D deficiency, elevated creatine kinase or ESR)
* If diabetic AND on sulfonylureas (like glipizide, glimepiride, glyburide), SGLT2 inhibitors (like dapagliflozin and empagliflozin), or insulin
* Undergoing treatment with any medications that affect bone turnover, including the following:

  * adrenocorticosteroids (> 3 months at any time or > 10 days within the previous yr), anticonvulsant therapy (within the previous year),
  * pharmacological doses of thyroid hormone (causing decline of thyroid stimulating hormone below normal),
  * calcium supplementation of > 1200 mg/d (within the preceding 3 months),
  * bisphosphonates (within the past 3 yrs),
  * denosumab,
  * estrogen (E) therapy or treatment with a selective E receptor modulator, or teriparatide (within the past yr).
* Subjects with a fracture within the past year
* Subjects taking potentially senolytic agents within the last year: Fisetin, Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax
* Subjects currently taking drugs that induce cellular senescence: alkylating agents, anthracyclines, platins, other chemotherapy
* QTc >450 msec
* Inability to provide informed consent
* Total bilirubin >2X upper limit
* Inability to tolerate oral medication
* eGFR < 15 ml/ min/ 1.73 m2
* Subjects on therapeutic doses of anticoagulants (e.g., warfarin, heparin, low molecular weight heparin, factor Xa inhibitors, etc.)
* Subjects taking the following antimicrobial agents: Aminoglycosides, Azole antifungals (fluconazole, miconazole, voriconazole, itraconazole), Macrolides (clarithromycin, erythromycin), Antivirals (nelfinavir, indinavir, saquinavir, ritonavir, elbasvir/grazoprevir), Rifampin
* Subjects taking proton pump inhibitors who are unable or unwilling to reduce or hold therapy prior to and during the 2-day Fisetin dosing
* Subjects taking the following other drugs if they cannot be held for at least 2 days before and during administration of Fisetin: digoxin, lithium, all statins, repaglidine, bosentan, gemfibrozil, olmesartan, enalapril, valsartan, methotrexate, corticosteroids, thyroid hormones, eluxadoline, eltrombopag, nitroglycerin, pioglitazone, glyburide, enzalutamide, ezetimibe, colchicine, imatinib, cyclosporine, tacolimus, sirolimus, carbamazepine, flecainide, phenytoin, phenobarbital, rifampicin, theophylline, warfarin, heparin, full dose ASA, clopidogrel, celecoxib, desipramine, thioridazine, venlafaxine, tizanidine, atomoxetine, voriconazole, citalopram, diazepam, escitalopram, propranolol, clozapine, cyclobenzaprine, mexiletine, olanzapine, ondansetron, riluzole
* In order to ensure vitamin D sufficiency, we will also exclude subjects with serum 25-hydroxyvitamin D levels of < 20 ng/ml.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2018-02-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Improved 6 minute walk | One Month
  Improved gait speed

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Pignolo, MD, PhD, Principal Investigator — Mayo Clinic; Sundeep Khosla, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No